CLINICAL TRIAL: NCT06699589
Title: Old School Hip Hop: Parent Follow-Up & Spanish Speakers Inclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, James M Noble, MD, MS, CPH, FAAN, Principal Investigator, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAR5473 - non-R01
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Dementia
Keywords: dementia; schools; nutrition; health education
MeSH Terms: conditions — Alzheimer Disease; Dementia; Health Education | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): School population without the Old SCHOOL Hip-Hop program, but with the My Plate program.
  Interventions: Behavioral: My Plate (Nutrition Education)
- Intervention (Experimental): School population with the Old SCHOOL Hip-Hop program.
  Interventions: Behavioral: Old SCHOOL Hip-Hop (Dementia Education)

INTERVENTIONS:
Behavioral: Old SCHOOL Hip-Hop (Dementia Education) — A school-based intervention called "Old S.C.H.O.O.L. Hip-Hop" (OSHH) or Seniors Can Have Optimal aging and Ongoing Longevity, to educate 4th and 5th grade students (ages 9-11y) about key dementia signs and symptoms, basic pathophysiology of Alzheimer disease, and the importance of early recognition, care-seeking behavior, and preventative measures (lifelong healthy lifestyle decisions). The intervention is delivered in a classroom or school auditorium setting, using an innovative, modular, multimedia program and home-based activities, to increase parental and family dementia literacy.
  Arms: Intervention
Behavioral: My Plate (Nutrition Education) — The program selected for the control arm, "My Plate," will address nutrition, physical activity, and obesity education. This program was selected because nutrition, physical activity, and wellness programs are now being incorporated into New York City public school curriculums as part of a legislative directive. Trained facilitators will conduct "My Plate" as an entry point for the USDA's My Plate nutrition program. Students will learn about My Plate across the 3-day one-hour-a-day program.
  Arms: Control

SUMMARY:
These are the exploratory aims of the original trial cohort study "Old School Hip Hop RCT (AAAR5473)," which recruited 783 parents.

1. Continued follow-up of these families to learn more about the durability of the program through similar assessments to those used during the pre-specified 3-month initial study timeframe - aiming to understand participant knowledge and personal experiences with family members or friends affected by Alzheimer's Disease (AD).
2. Further examining the degree of comfort with dementia, as measured by a simplified version of the Dementia Attitudes Scale (DAS) focused on observable behaviors in children by their parents - aiming to understand the extent of stigmatization of dementia in communities served by this program, and if the trial impacted evidence of stigma.
3. Enrolling up to 75 parents who primarily spoke Spanish who were originally contacted in the RCT but were not eligible for completion of the original round of surveys given that all study materials were in English. This approach aims to better understand the impact of the program and Alzheimer disease on these families.

Hypothesis 1: For the delayed follow-up with parents, the investigator anticipates that those with high dementia literacy or the largest dementia literacy improvement would sustain knowledge over 15-month period.

Hypothesis 2: Children who received the intervention arm of the trial, who also have regular contact with a close friend or family member with dementia, will demonstrate positive dementia attitudes relative to students in the control arm.

Hypothesis 3: Semi-structured interviews with Spanish speaking families will help program capacity to better serve the population and improve involvement in AD care and research.

DETAILED DESCRIPTION:
The goal of the R01 study is to educate children and thereby parents/guardians on health education content through live educators, music, and videos. The study curriculum focuses on healthy aging vs Dementia/Alzheimer's Disease (AD), nutrition, and overall health. The investigator wishes to learn if children are able to absorb these health topics and share what they learn with their parents/guardians. That part of the program has been completed with students. This non-R01 portion of the study is designed to look at the long-term effect of the program, how it may have affected Spanish speaking families that were not approached during the first portion.

ELIGIBILITY:
Inclusion Criteria:

* Parent that participated in the OSHH Trial
* Parent that expressed interest in participating, but originally excluded from OSHH Trial due to language barrier

Exclusion Criteria:

* Did not have a participating child in OSHH Trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Delayed Dementia Symptom and Response Knowledge Assessment Score | From 15 to 48 months post baseline data collection
  An instrument with multiple choice questions to assess knowledge of recognition of key signs/symptoms and ability to formulate the correct action plan in response to recognizing dementia. Parents were asked knowledge questions at three timepoints in main trial. This additional fourth time point would capture any changes in delayed knowledge retention (starting at 15-Months post baseline data collection).
Spanish Dementia Symptom and Response Knowledge Assessment Score (Spanish Speaking Parents) | From 2.5 to 6 years post student baseline collection
  Spanish Translated instrument with multiple choice questions to assess knowledge of recognition of key signs/symptoms and ability to formulate the correct action plan in response to recognizing dementia.

SECONDARY OUTCOMES:
Spanish Parent Semi-Structured Interview | From 2.5 to 6 years post student baseline collection
  Spanish Speaking parents were ineligible to complete baseline surveys related to language barriers in earlier program phase materials. This semi-structured interview aims to learn how to better serve this population when it comes to dementia education and research.
Adapted Dementia Attitude Scale for Children & Parents | From 15 to 48 months post baseline data collection
  An adapted instrument with multiple choice questions to assess parent and child dementia attitudes (comfort/stigma) post-program. At least 15 up to 48 months post baseline data collection.
Spanish Adapted Dementia Attitude Scale for Children & Parents (Spanish Speaking Parents) | From 2.5 to 6 years post student baseline collection
  A translated adapted instrument with multiple choice questions to assess parent and child dementia attitudes (comfort/stigma).

CONTACTS AND LOCATIONS:
Overall Officials: James M Noble, MD, Principal Investigator — Associate Professor, Taub Institute, Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No